CLINICAL TRIAL: NCT03703375
Title: Randomized Phase 3 Study Evaluation the Efficacy and Safety of Oral Azacitidine(CC-486) Compared to Investigator's Choice Therapy in Patients With Relapsed or Refractory Angioimmunoblastic T Cell Lymphoma
Brief Title: Efficacy and Safety of Oral Azacitidine (CC-486) Compared to Investigator's Choice Therapy in Patients With Relapsed or Refractory Angioimmunoblastic T Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OA-CL-LYM-LYSARC-13134C; U1111-1220-8294 (Registry Identifier: WHO)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, T-Cell
Keywords: CC-486; Azacitidine; Angioimmunoblastic; T Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma | interventions — Azacitidine; cc-486; romidepsin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Administration of Oral Azacitidine (CC-486) (Experimental): Oral azacytidine 300 mg during 14 first days of 28-days cycle for European (EU) patients, Oral azacytidine 200 mg during 14 first days of 28-days cycle for Asian patients (Treatment until progression, patient decision or toxicity)
  Interventions: Drug: Azacitidine
- Investigator's choice therapy - Romidepsin (Active Comparator): Romidepsin 14mg/m2 on days 1, 8 and 15 of a 28-days cycle (Treatment until progression, patient decision or toxicity)
  Interventions: Drug: Romidepsin
- Investigator's choice therapy - Gemcitabine (Active Comparator): Gemcitabine 1000mg/m2 on days 1, 8 and 15 of a 28-days cycle (during 6 cycles)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine
  Other Names: CC-486
  Arms: Administration of Oral Azacitidine (CC-486)
Drug: Romidepsin — Romidepsin
  Arms: Investigator's choice therapy - Romidepsin
Drug: Gemcitabine — Gemcitabine
  Arms: Investigator's choice therapy - Gemcitabine

SUMMARY:
This study is a multicentric, open-label, randomized phase 3 trial. The study will be conducted in select countries in Europe and South Korea sponsored by LYSARC and in Japan sponsored by Celgene. There will be a combined enrollment target of 86 randomized patients, with approximately 14 randomized patients from Japan.

The enrollment to the randomized study will start at European sites in parallel to a safety run-in part in Japan. A safety run-in will be conducted to confirm the tolerability of oral azacitidine at doses of 100 mg and 200 mg QD in Asian patients. Once oral azacitidine at 200 mg QD is confirmed as tolerable, Asian patients from Japan and South Korea will start to be randomized into the main study. Additional patients (non-randomized) are anticipated to enroll to the safety run-in.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted.
3. Patient is willing and able to adhere to the study visit schedule and other protocol requirements
4. Patient had local diagnosed peripheral T cell lymphoma (PTCL) with T-follicular helper (TFH) phenotype according to the criteria of the latest WHO classification based on a surgical lymph node biopsy or needle core biopsy including any one of

   * Angioimmunoblastic T cell lymphoma (AITL)
   * Follicular T cell lymphoma
   * Nodal peripheral T-cell lymphoma with TFH phenotype There should be a documented expression of minimum two TFH markers among this panel of markers: CD10, CXCL13, PD1, ICOS and BCL6 by the tumoral cells by immunohistochemistry. Biopsy at relapse or progression is not mandatory, but highly encouraged on a surgical or needle core biopsy, and diagnostic tissue should be available for central pathology review and for ancillary molecular studies.

   Local pathology report should be reviewed by the sponsor's medical monitor prior to enrollment.
5. ECOG performance status 0 to 3
6. Relapsed (after partial or complete response) or refractory AITL after at least one line of systemic therapy (there is no mandatory resting period after the previous treatment as long as the biochemistry and hematology labs meet the inclusion criteria as below.)
7. Meet the following lab criteria:

   * ANC ≥ 1,5 x 109/L (≥ 1 x 109/L if BM involvement by lymphoma)
   * Platelet ≥ 75 x 109/L (≥ 50 x 109/L if BM involvement by lymphoma)
   * Hemoglobin ≥ 8 g/dL.
8. Anticipated life expectancy at least 3 months
9. At least one measurable lesion on CT that is greater than 1.5 cm in the longest diameter for nodal lesions and greater than 1.0 cm in the longest diameter for extranodal lesions. The lesion must be measurable in two perpendicular dimensions. Patients with only cutaneous disease will be excluded.
10. Female patient of childbearing potential (FCBP) may participate, providing she meets the following conditions:

    Have two negative pregnancy tests as verified by the investigator prior to starting study treatment: serum pregnancy test at Screening and negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting treatment with study treatment (Cycle 1 Day 1). She must agree to ongoing pregnancy testing during the study (before beginning each subsequent cycle of treatment), and 28 days after the last study drug administration. This applies even if the patient practices complete abstinence from heterosexual contact.

    Agrees to practice true abstinence (which must be reviewed monthly and source documented) or agrees to the use of highly effective methods of contraception from 28 days prior to starting study treatment, and must agree to continue using such precautions during study treatment (including dose interruptions) and for up to 6 months after the last study drug administration. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptomthermal, post ovulation methods) and withdrawal are not acceptable methods of contraception. Cessation of contraception after this point should be discussed with a responsible physician.

    Agrees to abstain from breastfeeding during study participation and for at least 6 months after the last study drug administration.

    A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).
11. Male patient must either practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agrees to avoid fathering a child, to use highly effective methods of contraception, male condom plus spermicide during sexual contact with a pregnant female or a female of childbearing potential (even if he has undergone a successful vasectomy), from starting dose of IP (cycle 1 Day 1), including dose interruptions through 6 months after receipt of the last study drug administration.

    Furthermore, male patient must agree to not give semen or sperm during study drug therapy and for a period of 1 year after end of study drug therapy.
12. For EU countries, patient covered by a social security system

Exclusion Criteria:

1. Clinical evidence of central nervous system(CNS) involvement by lymphoma. Patients with suspicion of CNS involvement must undergo neurologic evaluation and CT/MRI of head and lumbar puncture to exclude CNS disease.
2. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision)
3. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
4. Known Human Immunodeficiency Virus (HIV) or Hepatitis C Virus (HCV) infection, or evidence of active Hepatitis B Virus (HBV) infection defined as:

   * HBs Ag positive
   * HBs Ag negative, anti-HBs antibody positive and/or anti-HBc antibody positive with detectable viral DNA
5. Impaired renal function (calculated MDRD or Cockcroft-Gault Creatinine Clearance < 30 ml/min) or impaired liver function tests (Serum total bilirubin level > 2.0 mg/dl [34 μmol/L] (except in case of Gilbert's Syndrome, or documented liver or pancreatic involvement by lymphoma), Serum transaminases (AST or ALT) > 3 upper normal limits) unless they are related to the lymphoma.
6. Active malignancy other than the one treated in this research. Prior history of malignancies, other than low risk MDS or CMML (with less than 5% blasts in bone marrow), unless the patient has been free of the disease for ≥ 3 years. However, patients with the following history/concurrent conditions are allowed:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histologic finding of prostate cancer (T1a or T1b) using the tumor, nodes, metastasis [TNM] clinical staging system
7. Treatment with any investigational drug within 5 half-lives before planned first cycle of study treatment and during the study. Ongoing medically significant adverse events from previous treatment, regardless of the time period.
8. Prior exposure to azacitidine and/ or any other demethylating agent (eg, decitabine)
9. Prior exposure to planned study treatment investigator's choice therapy (eg, prior exposure to gemcitabine is an exclusion if gemcitabine is the investigator's choice therapy prior to randomization)
10. Concurrent use of corticosteroids unless the patient is on a stable or decreasing dose for ≥ 1 week prior to informed consent form signature
11. Knowing or suspected hypersensitivity to active substance or to any of the excipients.
12. Pregnant, planning to become pregnant, or lactating woman
13. Candidate for hematopoietic stem cell transplantation
14. History of active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the oral azacitidine and/or predispose the patient to an increased risk of gastrointestinal toxicity per investigator's decision. Any condition causing inability to swallow tablets.
15. Significant active cardiac disease within the previous 6 months, including:

    * New York Heart Association (NYHA) class IV congestive heart failure
    * Unstable angina or angina requiring surgical or medical intervention; and/or
    * Myocardial infarction
16. Person deprived of his/her liberty by a judicial or administrative decision
17. Adult person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Japan (12):
  - Local Institution - 41822, Sapporo, Hokkaido
  - Local Institution - 41922, Okayama, Okayama-ken
  - Local Institution - 41722, Sayama, Osaka
  - Local Institution - 41422, Hidaka, Saitama-Pref
  - Local Institution - 40722, Chuo-ku, Tokyo
  - Local Institution - 40222, Koto-ku, Tokyo
  - Local Institution - 40922, Fukuoka
  - Local Institution - 40122, Isehara City, Kanagawa
  - Local Institution - 41522, Kashiwa
  - Local Institution - 41622, Nagoya
  - Local Institution - 41222, Sendai
  - Local Institution - 41322, Tsukuba

REFERENCES:
- [Derived] Dupuis J, Bachy E, Morschhauser F, Cartron G, Fukuhara N, Daguindau N, Casasnovas RO, Snauwaert S, Gressin R, Fox CP, d'Amore FA, Staber PB, Tournilhac O, Bouabdallah K, Thieblemont C, Andre M, Rai S, Ennishi D, Gkasiamis A, Nishio M, Fornecker LM, Delfau-Larue MH, Sako N, Mule S, de Leval L, Gaulard P, Tsukasaki K, Lemonnier F. Oral azacitidine compared with standard therapy in patients with relapsed or refractory follicular helper T-cell lymphoma (ORACLE): an open-label randomised, phase 3 study. Lancet Haematol. 2024 Jun;11(6):e406-e414. doi: 10.1016/S2352-3026(24)00102-9. PMID 38796193
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 participants were enrolled in the study. 86 participants received study treatment in the main study and 7 participants received doses in the safety run-in to monitor for dose limiting toxicities (DLTs). The safety run-in participants are pre-specified to be excluded from the analysis from primary and secondary outcome measures.
Groups:
- Oral Azacitidine: Participants received either safety run-in treatment or study treatment. In the safety run-in, participants received either 100 mg or 200 mg daily of oral azacitidine for 14 days in a 28-day schedule and observed for dose limiting toxicities (DLT). Study treatment was either 300 mg daily for 14 days of 28-day cycle or 200 mg daily for 14 days of 28-day cycle (Japanese participants). Oral azacitidine was self-administered on the first 14 days of each 28-day treatment cycle, unless there was a schedule modification due to disease progression, participant decision or unacceptable toxicity.
- Investigators Choice Therapy - Romidepsin: Single-agent Investigator's Choice Therapy - Romidepsin. Participants will receive treatment on a 28 day cycle with 14 mg/m2 administered on days 1, 8, and 15 of each cycle
- Investigators Choice Therapy - Bendamustine: Single-agent Investigator's Choice Therapy - Bendamustine. Participants will receive treatment on a 21-day cycle with 120 mg/m2 administered on days 1 and 2 of each cycle
- Investigators Choice Therapy - Gemcitabine: Single-agent Investigator's Choice Therapy - Gemcitabine. Participants will receive treatment on a 28-day cycle with 1000 mg/m2 (Japanese participants) or 1200 mg/m2 (EU participants) administered on days 1, 8, and 15 of each cycle.
Period: Pre-Randomization (Safety Run-In)
Arm/Group | Oral Azacitidine | Investigators Choice Therapy - Romidepsin | Investigators Choice Therapy - Bendamustine | Investigators Choice Therapy - Gemcitabine
Started | 7 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomization Period
Arm/Group | Oral Azacitidine | Investigators Choice Therapy - Romidepsin | Investigators Choice Therapy - Bendamustine | Investigators Choice Therapy - Gemcitabine
Started | 49 | 4 | 16 | 24
Safety Run-In | 7 | 0 | 0 | 0
Completed (Completed = ongoing to treatment period) | 42 | 4 | 16 | 23
Not Completed | 7 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Completed safety run-in treatment | 7 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Oral Azacitidine | Investigators Choice Therapy - Romidepsin | Investigators Choice Therapy - Bendamustine | Investigators Choice Therapy - Gemcitabine
Started | 42 | 4 | 16 | 23
Completed (Completed=ongoing treatment) | 0 | 0 | 4 | 5
Not Completed | 42 | 4 | 12 | 18
Not completed — Other Reasons | 0 | 1 | 0 | 3
Not completed — Consent Withdrawal | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 1 | 2
Not completed — Toxicity of Study Treatment | 2 | 0 | 4 | 1
Not completed — Progression | 32 | 1 | 7 | 11
Not completed — Completed treatment | 7 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Azacitidine | Investigators Choice Therapy - Romidepsin | Investigators Choice Therapy - Bendamustine | Investigators Choice Therapy - Gemcitabine | Total
Number analyzed (Participants) | 49 | 4 | 16 | 24 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (9.28) | 67.0 (7.16) | 60.8 (9.90) | 69.4 (10.80) | 67.8 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 1 | 6 | 9 | 38
  Male | 27 | 3 | 10 | 15 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data was not collected
Region of Enrollment [Count of Participants; unit: Participants]
  Asia | 15 | 4 | 0 | 3 | 22
  Europe | 34 | 0 | 16 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Local Assessment
Description: PFS is defined as the time from randomization into the study to the first observation of documented disease progression (local assessment using Lugano Response Criteria 2014) or death due to any cause, whichever occurs first. If a participant has not progressed or died, PFS will be censored at the time of last visit with adequate assessment. C2 censoring rules were used per US FDA guidance 2015. Progression will be determined as per Response criteria for lymphoma: Lugano classification.
Time Frame: From randomization up to documented disease progression or death, whichever occurs first (up to approximately 15 months)
Population: Intent-to-Treat (ITT) population: all participants having signed their informed consent and who are randomized into the trial, regardless of they received study treatment or not.
  This endpoint is a pre-specified analysis intended to combine all investigator's choice participants, regardless of the specific investigator's choice treatment that was administered.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine): Single-agent Investigator's Choice Therapy - Romidepsin. Participants will receive treatment on a 28 day cycle with 14 mg/m2 administered on days 1, 8, and 15 of each cycle
  Single-agent Investigator's Choice Therapy - Bendamustine. Participants will receive treatment on a 21-day cycle with 120 mg/m2 administered on days 1 and 2 of each cycle
  Single-agent Investigator's Choice Therapy - Gemcitabine. Participants will receive treatment on a 28-day cycle with 1000 mg/m2 (Japanese participants) or 1200 mg/m2 (EU participants) administered on days 1, 8, and 15 of each cycle.
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 42 | 44
Months | 5.6 [2.66 to 7.26] | 2.8 [1.87 to 4.83]
Statistical Analysis 1: Comparison: Oral Azacitidine vs Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine); Test type: Superiority; p = 0.0541, Stratified Cox; Stratified Cox proportional hazards model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.41 to 1.09]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. OS was censored at the last date that the participant was known to be alive.
Time Frame: From randomization up to the date of death or date last known alive (up to approximately 27 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 42 | 44
Months | 18.4 [12.88 to 31.47] | 10.3 [4.24 to 13.50]
Statistical Analysis 1: Comparison: Oral Azacitidine vs Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine); Test type: Superiority; p = 0.0166, Efron; Stratified Cox proportional hazards model; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.32 to 0.96]

3. Secondary Outcome: Progression Free Survival (PFS) Based on IRC Assessment
Description: PFS based on Independant Review Committee (IRC) is defined as the time from randomization into the study to the first observation of documented disease progression (reviewed assessment by IRC using Lugano Response Criteria 2014) or death due to any cause. If a patient has not progressed or died, PFS will be censored at the time of last visit with adequate assessment per FDA's guidance 2015 Table C2. Progression will be determined as per Response criteria for lymphoma: Lugano classification.
Time Frame: From randomization up to documented disease progression or death, whichever occurs first (up to approximately 37 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 42 | 44
Months | 4.2 [2.66 to 5.88] | 3.2 [2.10 to 4.83]
Statistical Analysis 1: Comparison: Oral Azacitidine vs Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine); Test type: Superiority; p = 0.2139, Stratified Cox; Stratified Cox proportional hazards model; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.51 to 1.33]

4. Secondary Outcome: Overall Response Rates (ORR)
Description: Overall response rates are the percentage of complete response (CR) and partial response (PR) per local assessment. Assessment of response will be based on Lugano Response Criteria 2014 for the radiologic response (CT based), the metabolic response (PET-CT based) and the best response between radiologic and metabolic response. Measurements occurred after Cycle 3, after Cycle 6, and at permanent treatment discontinuation. PR is defined as Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size and ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites. CR is defined as target nodes/nodal masses regressed to ≤ 1.5 cm in LDi, no extralymphatic sites of disease, and Score 1, 2, or 3 with or without a residual mass on the 5 Point Scale. The Lugano 5-point scale is 1, no uptake above background; 2, uptake mediastinum; 3, uptake mediastinum but liver; 4, uptake moderately liver; 5, uptake markedly higher than liver and/or new lesions.
Time Frame: Response rate will be measured after Cycle 3, after Cycle 6 (up to approximately 5.5 months)
Population: CR and PR responders in Intent-to-Treat population.
  This endpoint is a pre-specified analysis intended to combine all investigator's choice participants, regardless of the specific investigator's choice treatment that was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 14 | 19
Percentage of participants
  Cycle 3 | 33.3 [19.6 to 49.5] | 43.2 [28.3 to 59.0]
  Cycle 6: number analyzed (Participants) | 13 | 10
  Cycle 6 | 31.0 [17.6 to 47.1] | 22.7 [11.5 to 37.8]

5. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate is the percentage of CR (complete metabolic response or CT-based CR) per local assessment before receiving any subsequent anti-lymphoma therapy. Assessment will be based on Lugano Response Criteria 2014 for the radiologic response (CT based), the metabolic response (PET-CT based) and best response between radiologic and metabolic response. Measurements occurred after Cycle 3, Cycle 6, and treatment discontinuation. PR is defined as Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size and ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites. CR is defined as target nodes/nodal masses regressed to ≤ 1.5 cm in LDi, no extralymphatic sites of disease, and Score 1, 2, or 3 with or without a residual mass. The Lugano 5-point scale is 1, no uptake above background; 2, uptake mediastinum; 3, uptake mediastinum but liver; 4, uptake moderately liver; 5, uptake markedly higher than liver and/or new lesions.
Time Frame: Response rate will be measured after Cycle 3, after Cycle 6 (up to approximately 5.5 months)
Population: CR and PR responders in Intent-to-Treat population
  This endpoint is a pre-specified analysis intended to combine all investigator's choice participants, regardless of the specific investigator's choice treatment that was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 5 | 10
Percentage of participants
  Cycle 3 | 11.9 [4.0 to 25.6] | 22.7 [11.5 to 37.8]
  Cycle 6: number analyzed (Participants) | 5 | 7
  Cycle 6 | 11.9 [4.0 to 25.6] | 15.9 [6.6 to 30.1]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from attainment of complete response (CR) or partial response (PR) per local assessment to the date of first documented disease progression, relapse (local assessment) or death from any cause. Participants alive and free of progression will be censored at their last visit with adequate assessment.CR: complete metabolic response or computed tomography (CT)-based CR; PR: partial metabolic response or CT-based PR before subsequent anti-lymphoma therapy.
Time Frame: From randomization to the date of first documented disease progression, relapse (local assessment) or death from any cause (up to approximately 27 months)
Population: CR or PR responders in Intent-to-Treat population
  This endpoint is a pre-specified analysis intended to combine all investigator's choice participants, regardless of the specific investigator's choice treatment that was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 17 | 19
Percentage of participants | 10.4 [2.56 to NA] — Upper limit not calculated due to insufficient number of events | 3.4 [2.00 to NA] — Upper limit not calculated due to insufficient number of events

7. Secondary Outcome: Time to Response (TTR)
Description: Time to response is defined as the time from randomization to the date of attainment of complete response (CR) or partial response (PR) per local assessment until end of treatment. If a participant is not responder, time to response will be censored at the time of last visit with adequate assessment. CR: complete metabolic response or computed tomography (CT)-based CR; PR: partial metabolic response or CT-based PR before subsequent anti-lymphoma therapy.
Time Frame: From randomization to the date of attainment of complete response (CR) or partial response (PR) until end of treatment (up to approximately 37 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 17 | 19
Months | 3 [3 to 6] | 2.7 [1 to 4]

8. Secondary Outcome: Progression Free Survival 2 (PFS2) on Local Assessment
Description: PFS2 based on local assessment is defined as the time from randomization to objective tumor progression on next-line treatment or death from any cause. Participants without next-line therapy who did not die and participants who did not relapse or not die after next-line therapy will be censored at the last adequate tumor assessment date.
Time Frame: From randomization to objective tumor progression on next-line treatment or death from any cause (up to approximately 27 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine | Investigators Choice Therapy Combined (Romidepsin, Bendamustine, Gemcitabine)
Number analyzed (Participants) | 42 | 44
Months | 11.0 [6.44 to 18.89] | 6.7 [3.52 to 9.56]

9. Secondary Outcome: Mean Change in Minimal Important Differences (MIDs) of the EORTC QLQ-C30 Health-related Quality-of-Life Domain Scores
Description: The minimal important difference (MID) is the size of difference in Quality-of-Life score that is considered relevant (i.e. warranting a change in treatment or examinations). The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQC30) subscale values are the lower threshold for MID over time, based on within-group mean change. QLQ-C30 has 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain), a global health status / quality of life (QoL) scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). Each scale was scored on a range from 0 to 100. Higher scores represent a higher response level. Note that a high score for global health status or for a functional scale represents a high or healthy level of functioning, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time Frame: At baseline and on Day 1 of each cycle up to treatment discontinuation (up to approximately 27 months)
Reporting Status: Not Posted, anticipated posting 2025-02

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 37 months). SAEs and Other AEs were assessed from first dose to 28 days following last dose (up to approximately 38 months)
Groups:
- Oral Azacitidine: 200 mg: Participants received 200 mg daily for 14 days of 28-day cycle (Japanese participants). Oral azacitidine was self-administered on the first 14 days of each 28-day treatment cycle, unless there was a schedule modification due to disease progression, subject decision or unacceptable toxicity.
- Oral Azacitidine: 300 mg: Participants received 300 mg daily for 14 days of 28-day cycle. Oral azacitidine was self-administered on the first 14 days of each 28-day treatment cycle, unless there was a schedule modification due to disease progression, subject decision or unacceptable toxicity.
- Investigators Choice Therapy - Gemcitabine: 1000 mg/m2: Single-agent Investigator's Choice Therapy - Gemcitabine. Participants will receive treatment on a 28-day cycle with 1000 mg/m2 administered on days 1, 8, and 15 of each cycle
- Investigators Choice Therapy - Gemcitabine: 1200 mg/m2: Single-agent Investigator's Choice Therapy - Gemcitabine. Participants will receive treatment on a 28-day cycle with 1200 mg/m2 administered on days 1, 8, and 15 of each cycle
- Safety Run-in Oral Azacitidine: 100 mg: In the safety run-in, participants received 100 mg daily of oral azacitidine for 14 days in a 28-day schedule and observed for dose limiting toxicities (DLT)
- Safety Run-in Oral Azacitidine: 200 mg: In the safety run-in, participants received 200 mg daily of oral azacitidine for 14 days in a 28-day schedule and observed for dose limiting toxicities (DLT)
Arm/Group | Oral Azacitidine: 200 mg | Oral Azacitidine: 300 mg | Investigators Choice Therapy - Romidepsin | Investigators Choice Therapy - Bendamustine | Investigators Choice Therapy - Gemcitabine: 1000 mg/m2 | Investigators Choice Therapy - Gemcitabine: 1200 mg/m2 | Safety Run-in Oral Azacitidine: 100 mg | Safety Run-in Oral Azacitidine: 200 mg
All-Cause Mortality (participants affected / at risk) | 6/8 | 20/34 | 1/4 | 13/16 | 3/3 | 14/21 | 1/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/8 | 9/34 | 2/4 | 8/16 | 0/3 | 9/20 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 7/8 | 33/34 | 4/4 | 16/16 | 3/3 | 19/20 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine: 200 mg (N=8) | Oral Azacitidine: 300 mg (N=34) | Investigators Choice Therapy - Romidepsin (N=4) | Investigators Choice Therapy - Bendamustine (N=16) | Investigators Choice Therapy - Gemcitabine: 1000 mg/m2 (N=3) | Investigators Choice Therapy - Gemcitabine: 1200 mg/m2 (N=20) | Safety Run-in Oral Azacitidine: 100 mg (N=3) | Safety Run-in Oral Azacitidine: 200 mg (N=3)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Clostridium colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis aspergillus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visceral leishmaniasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine: 200 mg (N=8) | Oral Azacitidine: 300 mg (N=34) | Investigators Choice Therapy - Romidepsin (N=4) | Investigators Choice Therapy - Bendamustine (N=16) | Investigators Choice Therapy - Gemcitabine: 1000 mg/m2 (N=3) | Investigators Choice Therapy - Gemcitabine: 1200 mg/m2 (N=20) | Safety Run-in Oral Azacitidine: 100 mg (N=3) | Safety Run-in Oral Azacitidine: 200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 | 10 | 1 | 2 | 1 | 9 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 15 | 3 | 14 | 3 | 15 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 15 | 3 | 9 | 2 | 11 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | 4 | 7 | 2 | 8 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 11 | 1 | 2 | 0 | 1 | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 9 | 1 | 1 | 0 | 5 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 17 | 2 | 5 | 0 | 6 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 14 | 1 | 2 | 0 | 1 | 1 | 3
Asthenia (General disorders) | 0 | 8 | 0 | 3 | 0 | 3 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 1 | 1 | 1 | 5 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 1 | 1 | 2 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT03703375/Prot_SAP_000.pdf